CLINICAL TRIAL: NCT03545451
Title: Neurofeedback Rehabilitation Based on Motor Imaging in Patients in the Immobilization Phase
Acronym: REMINARY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K170502J
Record Dates: First submitted 2018-04-05; First posted 2018-06-04 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-05

CONDITIONS: Healthy Subjects, Patients With Amyotrophic Lateral Sclerosis, Patients With Shoulder Surgery
Keywords: EEG, neurofeedback, fMRI, ALS, surgery, upper limbs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofeedback rehabilitation with videogames (Experimental): Neurofeedback rehabilitation with videogames
  Interventions: Device: Videogames

INTERVENTIONS:
Device: Videogames — Videogames

SUMMARY:
As the prevalence of motor impairment increases with age, the proportion of the population affected by physical limitations is likely to increase in the coming years, considering that one in three people will be over 60 in 2050 (compared to one in five in 2005, INSEE projections). The possibility of reducing recovery time and / or improving the improvement of motor deficits is today a public health issue. The possibility of developing new therapeutic tools using innovative motor imaging rehabilitation technologies is an opportunity to offer rehabilitation adapted to specific disorders, personalized in relation to the patient's performance, and in continuity with the therapist. In this research project, we will use the principle of neurofeedback rehabilitation (EEG) based on motor imaging with a brain-computer interface. Feedback will consist of therapeutic video games.Here, we will test the feasibility of such approach in 10 healthy subjects, 10 patients with amyotrophic lateral sclerosis and 10 patients with uppel shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

Common to the 3 populations concerned:

* patients or subjects of both sexes;
* age: 18-70 years;
* ability to give consent in writing;
* Health Insurance.

  a) SLA:
* patients with amyotrophic lateral sclerosis (defined according to the El Escorial criteria: possible, probable or definite), at the time of diagnosis;
* Percentage of forced vital capacity (FVC) ≥ 65% of the predicted value for age, gender and size.

  b) Patients after a shoulder trauma: patients with scheduled shoulder surgery. c) Healthy subjects.

Exclusion Criteria:

* Dementia (MMSE score <24/30)
* Pregnancy or patient not having effective contraception.
* Other neurological, psychiatric or orthopedic disease leading to a motor handicap or an inability to correctly realize the experimental paradigm: interfering with the evaluation of the movements of the upper limb, incapacity to realize the mental imagery of the movement.
* Visual impairment resulting in an inability to properly view the computer screen.
* History of epilepsy or active epilepsy.
* Contraindication to MRI: cardiac or neuronal simulator, ferromagnetic surgical clips, implants and metal objects, intraocular foreign bodies, claustrophobia
* Persons under guardianship, trusteeship or any other administrative or judicial measure of deprivation of rights and liberty
* Subject in the exclusion period of another interventional research or participating in any other interventional research or therapeutic trial
* Presence of another severe progressive pathology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Performance | week 1
  total displacement fo the avatar within the game

SECONDARY OUTCOMES:
electroencephalography activity | week 1, 2, 3, 4, 5 and 6
  amplitude of the oscillatory activity
functional brain MRI | week 1 and 6
  BOLD signal

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe Corvol, MD, PHD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière Paris, France, 75013
Locations (1):
- Hopital PITIE SALPETRIERE, Paris, France